CLINICAL TRIAL: NCT05332431
Title: Optical Coherence Tomography Findings in Patients With Different Types of Migraine
Brief Title: Optical Coherence Tomography Findings in Migraine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad El din Mahmoud Taher, Principal investigator, Resident doctor of Neurology, Assiut University
Other Study IDs: OCT in migraine
Record Dates: First submitted 2021-12-13; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Migraine: Patients diagnosed with migraine based on prespecified criteria according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3) established by established by the International Headache Society, for migraine with aura and migraine without aura, attending the neurology outpatient clinic, Assiut University.
  Interventions: Device: Optical coherence tomography (OCT)
- Control: Age and sex matched healthy control group (with the absence of any pathological headache and eye problems), will be recruited from the outpatient clinic for comparison.
  Interventions: Device: Optical coherence tomography (OCT)

INTERVENTIONS:
Device: Optical coherence tomography (OCT) — Patient with different types of migraine and age and sex matched control group will be subjected to OCT in the ophthalmology department in Assiut University Hospital to assess the following parameters:
  Optic nerve head parameters and retinal nerve fibre layer thickness and measuring macular thickness in migraine patients will be measured using optical coherence tomography (OCT) after pupillary dilatation. Retinal nerve fiber layer thickness included average thickness (360° measurement), temporal quadrant thickness (316-45°), superior quadrant thickness (46-135°), nasal quadrant thickness (136-225°) and inferior quadrant thickness (226-315°) will be measured by OCT.

SUMMARY:
This study aims to detect changes in RNFL thickness in patients with different types of migraine in comparison to healthy control. This will be accomplished by comparing the optic nerve head (ONH) parameters, RNFL thickness, and ocular perfusion pressure (OPP) in migraine patients with age and sex matched healthy control.

DETAILED DESCRIPTION:
Migraine is a complex, neurological disorder with a genetic basis . It a primary type of headache that characterized by moderate to severe intensity pain associated with fatigue, depression, hyperactivity, nausea, sensitivity to light or sound and other neurological symptoms . The international classification of headaches divides migraine into two main types: migraine without aura and migraine with aura.

It affects a large range of individuals, although it more commonly begins in the first few decades of life . According to World Health Organization data, migraine has become the third most common disease in the 21st century . In the meantime, migraine is one of the top ten causes of disability in the world . Based on the WHO reports, Atlas of Headache Disorders and Resources in the World 2011, migraine affects 11% of adults worldwide, and females have three times higher prevalence than males, and it is the leading cause of years lost due to disability in individuals aged 15 to 49 years. Migraine has generally increased in incidence worldwide in recent years, especially in developing countries, possibly with adverse lifestyle changes brought about by rapid urbanization in these regions.

There is no consensus on the pathogenesis of migraine, but it is generally accepted that migraine is caused by the combined involvement of nerves and blood vessels . Cortical spreading depression (CSD) has been known to play an important role in the pathogenesis of migraine, which can activate and sensitize the trigeminal vascular system (TGVS), then triggers migraine-associated neurological and vascular responses, and finally induces pain. There are four potential phases of migraine have been identified, including the premonitory phase, aura, headache, and the postdrome, and these are not necessarily linear in occurrence. A better comprehension of the underlying pathophysiology of these phases has led to, for the first time in history, new preventive treatments coming out tailored specifically to treat the mechanism of migraine.

Although migraine is a transient phenomenon of cerebral vasoconstriction, transitory and recurrent constriction of the retinal and ciliary arteries may cause ischemic damage to the optic nerve, retina, and choroid in patients with migraine . There is evidence that ganglion cell death in migraine patients may be secondary to alterations in the microcirculation of the optic nerve head or even in the quality of retinal perfusion Though brain and retina come from the same embryologic origin, retina provides a unique window into the nervous system because of having unmyelinated axons and a low concentration of glial cells. That is why retina is called "a relative vacuum" while studying neurons and axons and it can serve as a valuable surrogate marker of neurodegeneration and neuroprotection.

Optical coherence tomography (OCT) was developed as a noninvasive technique for acquiring in vivo cross-sectional images during the 1980s and 1990s . Over the last 20 years, OCT has been extensively applied by ophthalmologists to study ocular pathologies, but in these days, it is also being used by neurologists and was studied as a biomarker in various neurologic conditions.

There are many studies investigated the altered retinal nerve fiber layer (RNFL) thickness by using OCT in migraine patients but the findings were inconsistent. Some studies reported reduction of RNFL thickness in patient with migraine. While other studies reported normal thickness of RNFL and did not find any statistically significant change in RNFL thickness between different types of migraine and between migraine and control groups. The present study aims to detect changes in RNFL thickness in patients with different types of migraine in comparison to healthy control.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfill the criteria of case definition of migraine with aura and migraine without aura.
* Gender: both sexes are included.
* Willingness to participate in the study and to be subjected to the disease-related examinations and assessments.
* Willing and able to provide informed consent

Exclusion Criteria:

* Unable to give informed consent.
* History of chronic psychiatric or neurological disorder as patients with history of central nervous system disorders including brain tumours, infarction, epilepsy, Alzheimer's disease, and any type of headache except for migraine.
* Patients with known systemic diseases (such as diabetes mellitus and hypertension).
* Patients with known ophthalmic disorders, refractive error exceeding ± 3.0 diopters and had previously undergone any type of eye surgery. Those with optic disc anomaly, hazy media, and any retinal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients diagnosed with migraine based on prespecified criteria according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3) established by established by the International Headache Society, for migraine with aura and migraine without aura, attending the neurology outpatient clinic, Assiut University.
  2. Age and sex matched healthy control group (with the absence of any pathological headache and eye problems), will be recruited from the outpatient clinic for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in retinal nerve fiber layer thickness (RNFL) measured by OCT. | Baseline
  Patient with different types of migraine and age and sex matched control group will be subjected to OCT in the ophthalmology department in Assiut University Hospital to assess the following parameters:
  Optic nerve head parameters and retinal nerve fibre layer thickness and measuring macular thickness in migraine patients will be measured using optical coherence tomography (OCT) after pupillary dilatation. Retinal nerve fiber layer thickness included average thickness (360° measurement), temporal quadrant thickness (316-45°), superior quadrant thickness (46-135°), nasal quadrant thickness (136-225°) and inferior quadrant thickness (226-315°) will be measured by OCT.

SECONDARY OUTCOMES:
Correlations of OCT findings in patients with migraine with migraine severity. | Baseline
  Correlate the findings of OCT with the severity of the migraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qubty W, Patniyot I. Migraine Pathophysiology. Pediatr Neurol. 2020 Jun;107:1-6. doi: 10.1016/j.pediatrneurol.2019.12.014. Epub 2020 Feb 4. PMID 32192818
- [Background] Giffin NJ, Ruggiero L, Lipton RB, Silberstein SD, Tvedskov JF, Olesen J, Altman J, Goadsby PJ, Macrae A. Premonitory symptoms in migraine: an electronic diary study. Neurology. 2003 Mar 25;60(6):935-40. doi: 10.1212/01.wnl.0000052998.58526.a9. PMID 12654956
- [Background] Vecchia D, Pietrobon D. Migraine: a disorder of brain excitatory-inhibitory balance? Trends Neurosci. 2012 Aug;35(8):507-20. doi: 10.1016/j.tins.2012.04.007. Epub 2012 May 24. PMID 22633369
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Barnett R. Migraine. Lancet. 2019 Nov 23;394(10212):1897. doi: 10.1016/S0140-6736(19)32763-1. Epub 2019 Nov 21. No abstract available. PMID 31982043
- [Background] Buse DC, Silberstein SD, Manack AN, Papapetropoulos S, Lipton RB. Psychiatric comorbidities of episodic and chronic migraine. J Neurol. 2013 Aug;260(8):1960-9. doi: 10.1007/s00415-012-6725-x. Epub 2012 Nov 7. PMID 23132299
- [Background] Wang SJ, Chen PK, Fuh JL. Comorbidities of migraine. Front Neurol. 2010 Aug 23;1:16. doi: 10.3389/fneur.2010.00016. eCollection 2010. PMID 21188255
- [Background] Michael NDB, Hussein A, Abd Halim S, Ab Hamid SA. Evaluation of Optic Nerve Head Parameters, Retinal Nerve Fiber Layer Thickness, and Ocular Perfusion Pressure in Migraine Patients. Cureus. 2019 May 4;11(5):e4599. doi: 10.7759/cureus.4599. PMID 31309023
- [Background] Steiner TJ, Stovner LJ, Vos T, Jensen R, Katsarava Z. Migraine is first cause of disability in under 50s: will health politicians now take notice? J Headache Pain. 2018 Feb 21;19(1):17. doi: 10.1186/s10194-018-0846-2. No abstract available. PMID 29468450
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Woldeamanuel YW, Cowan RP. Migraine affects 1 in 10 people worldwide featuring recent rise: A systematic review and meta-analysis of community-based studies involving 6 million participants. J Neurol Sci. 2017 Jan 15;372:307-315. doi: 10.1016/j.jns.2016.11.071. Epub 2016 Dec 3. PMID 28017235
- [Background] Burstein R, Noseda R, Borsook D. Migraine: multiple processes, complex pathophysiology. J Neurosci. 2015 Apr 29;35(17):6619-29. doi: 10.1523/JNEUROSCI.0373-15.2015. PMID 25926442
- [Background] Goadsby PJ, Charbit AR, Andreou AP, Akerman S, Holland PR. Neurobiology of migraine. Neuroscience. 2009 Jun 30;161(2):327-41. doi: 10.1016/j.neuroscience.2009.03.019. Epub 2009 Mar 19. PMID 19303917
- [Background] Cutrer FM. Pathophysiology of migraine. Semin Neurol. 2010 Apr;30(2):120-30. doi: 10.1055/s-0030-1249222. Epub 2010 Mar 29. PMID 20352582
- [Background] Ayata C. Cortical spreading depression triggers migraine attack: pro. Headache. 2010 Apr;50(4):725-30. doi: 10.1111/j.1526-4610.2010.01647.x. PMID 20456160
- [Background] Gipponi S, Scaroni N, Venturelli E, Forbice E, Rao R, Liberini P, Padovani A, Semeraro F. Reduction in retinal nerve fiber layer thickness in migraine patients. Neurol Sci. 2013 Jun;34(6):841-5. doi: 10.1007/s10072-012-1103-0. Epub 2012 Apr 26. PMID 22535509
- [Background] Zengin MO, Elmas Z, Cinar E, Kucukerdonmez C. Choroidal thickness changes in patients with migraine. Acta Neurol Belg. 2015 Mar;115(1):33-7. doi: 10.1007/s13760-014-0301-3. Epub 2014 May 8. PMID 24806667
- [Background] Ascaso FJ, Marco S, Mateo J, Martinez M, Esteban O, Grzybowski A. Optical Coherence Tomography in Patients with Chronic Migraine: Literature Review and Update. Front Neurol. 2017 Dec 13;8:684. doi: 10.3389/fneur.2017.00684. eCollection 2017. PMID 29321760
- [Background] Martinez A, Proupim N, Sanchez M. Retinal nerve fibre layer thickness measurements using optical coherence tomography in migraine patients. Br J Ophthalmol. 2008 Aug;92(8):1069-75. doi: 10.1136/bjo.2008.137471. Epub 2008 Jul 9. PMID 18614573
- [Background] Martinez A, Proupim N, Sanchez M. Scanning laser polarimetry with variable corneal compensation in migraine patients. Acta Ophthalmol. 2009 Nov;87(7):746-53. doi: 10.1111/j.1755-3768.2008.01356.x. PMID 18811640
- [Background] Greenberg BM, Frohman E. Optical coherence tomography as a potential readout in clinical trials. Ther Adv Neurol Disord. 2010 May;3(3):153-60. doi: 10.1177/1756285610368890. PMID 21179607
- [Background] Huang D, Swanson EA, Lin CP, Schuman JS, Stinson WG, Chang W, Hee MR, Flotte T, Gregory K, Puliafito CA, et al. Optical coherence tomography. Science. 1991 Nov 22;254(5035):1178-81. doi: 10.1126/science.1957169.
- [Background] Mokbul MI. Optical Coherence Tomography: Basic Concepts and Applications in Neuroscience Research. J Med Eng. 2017;2017:3409327. doi: 10.1155/2017/3409327. Epub 2017 Oct 29. PMID 29214158
- [Background] Lin X, Yi Z, Zhang X, Liu Q, Cai R, Chen C, Zhang H, Zhao P, Pan P. Retinal nerve fiber layer changes in migraine: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Aug 14;99(33):e21680. doi: 10.1097/MD.0000000000021680. PMID 32872037
- [Background] Bulboaca AE, Stanescu IC, Bolboaca SD, Bulboaca AC, Bodizs GI, Nicula CA. Retinal Nerve Fiber Layer Thickness and Oxidative Stress Parameters in Migraine Patients without Aura: A Pilot Study. Antioxidants (Basel). 2020 Jun 5;9(6):494. doi: 10.3390/antiox9060494. PMID 32516927
- [Background] Simsek IB, Aygun D, Yildiz S. Retinal Nerve Fibre Layer Thickness in Migraine Patients with or without Aura. Neuroophthalmology. 2014 Nov 24;39(1):17-21. doi: 10.3109/01658107.2014.968740. eCollection 2015 Feb. PMID 27928325
- [Background] Salman AG, Hamid MA, Mansour DE. Correlation of visual field defects and optical coherence tomography finding in migraine patients. Saudi J Ophthalmol. 2015 Jan-Mar;29(1):76-80. doi: 10.1016/j.sjopt.2014.06.008. Epub 2014 Jul 1. PMID 25859145
- [Background] Peng KP, Wang SJ. Migraine diagnosis: screening items, instruments, and scales. Acta Anaesthesiol Taiwan. 2012 Jun;50(2):69-73. doi: 10.1016/j.aat.2012.05.002. Epub 2012 Jun 19. PMID 22769861
- [Background] Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology. 2001;56(6 Suppl 1):S20-8. doi: 10.1212/wnl.56.suppl_1.s20. PMID 11294956